CLINICAL TRIAL: NCT02064023
Title: Comparison of Continuous Subcutaneous Insulin Infusion (CSII) With Multiple Daily Injections (MDI) for the Treatment of Pregestational Diabetes During Pregnancy
Brief Title: Comparison of Insulin Pump and MDI for Pregestational Diabetes During Pregnancy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Some sites withdrew because no contract with insulin pump supplier
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, David Thompson, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H12-02375
Record Dates: First submitted 2014-02-03; First posted 2014-02-17 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes; Pregnancy
Keywords: insulin pump; CSII; multiple daily injections; MDI; type 1 diabetes; type 2 diabetes; pregnancy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Infusion Systems

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- insulin pump (Experimental): subjects will use an insulin pump for the duration of the pregnancy. The intervention is that they will control their diabetes using an insulin pump
  Interventions: Device: insulin pump
- Multiple Daily Insulin injections (Active Comparator): subjects will continue their usual insulin treatment with multiple daily injections of sc insulin
  Interventions: Other: multiple daily insulin injection

INTERVENTIONS:
Device: insulin pump — subjects in the experimental arm will administer insulin using a pump
  Arms: insulin pump
Other: multiple daily insulin injection — Subjects will continue with usual insulin injections
  Arms: Multiple Daily Insulin injections

SUMMARY:
This study is investigating whether insulin treatment with the insulin pump or with multiple daily injections (MDI) gives better outcomes for mother and baby in pregnant women with pregestational diabetes. Participants will be randomized to use either the insulin pump or MDI.

DETAILED DESCRIPTION:
Primary outcome is a composite of Cesarian section, instrumental delivery, maternal hypertension, LGA infant, neonatal hypoglycemia or SCN admission.

ELIGIBILITY:
Inclusion Criteria:

* subjects are attending the Diabetes Pregnancy Clinic at participating hospitals
* have had type 1 or type 2 diabetes for at least one year
* are in the first trimester or are actively attempting pregnancy
* have a singleton pregnancy
* are receiving intensive insulin therapy
* are judged by clinic staff to be capable of using an insulin pump
* are age 19 or older
* are willing to adhere to the study protocol including monitoring blood glucose levels
* are willing to take folic acid before pregnancy and during the first trimester
* are willing to discontinue any medication contraindicated in pregnancy prior to conception
* weigh less than 100 kg (220 lb) prior to becoming pregnant
* use less than 100 units of insulin per day

Exclusion Criteria:

* current or previous use of an insulin pump
* use of fertility treatments
* have a multiple pregnancy
* have had children born with major birth defects
* have experienced stillbirth or multiple early pregnancy losses
* have significant diabetes complications or a serious medical issue

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12-04 (Actual); Study Completion 2015-12-04 (Actual)

PRIMARY OUTCOMES:
Composite obstetrical/perinatal endpoint consisting of specific elements (see description) | Up to 42 weeks
  Composite obstetrical/perinatal endpoint consisting of one or more of pre-eclampsia, primary caesarian section, pre-term delivery, spontaneous abortion, termination for congenital anomaly or chromosomal abnormality, perinatal mortality, large-for-gestational age, shoulder dystocia, birth injury, major congenital anomaly, neonatal hypoglycemia, jaundice requiring phototherapy, or admission to neonatal intensive care nursery.

SECONDARY OUTCOMES:
Mean maternal HbA1c during pregnancy | up to 42 weeks
  HbA1c will be measured at least every three months to provide information about overall glycemic control

OTHER OUTCOMES:
Number of episodes of severe hypoglycemia | up to 42 weeks
  Severe hypoglycemia is defined as capillary glucose < 3.3 mmol/L requiring the assistance of another person for treatment.

CONTACTS AND LOCATIONS:
Overall Officials: David M Thompson, MD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Jim Pattison Outpatient Care and Surgery Centre, Surrey, British Columbia
  - B.C. Women's Hospital, Vancouver, British Columbia